CLINICAL TRIAL: NCT02891876
Title: 3-months Success Rate of Direct Pulp Capping With Biodentine®
Acronym: CPDB
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: CPDB
Record Dates: First submitted 2016-08-30; First posted 2016-09-08 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Dental Pulp Capping
Keywords: direct pulp capping, biodentine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Biodentine® is a most recent material for direct pulp capping. The aim of this study is to determine the 3 months success rate (defined as clinical and radiographic successes together) of direct pulp capping realized with Biodentine®.

DETAILED DESCRIPTION:
Context : When a pulpal exposure happens on a vital tooth (without irreversible inflammation), direct pulp capping can be realized by using different biomaterials : CaOH2, MTA or Biodentine®. Biodentine® is the most recent material and its success rate for direct pulp capping is poorly documented.

Objective : The main aim of this study is to determine the 3 months success rate (defined as clinical and radiographic successes together) of direct pulp capping realized with Biodentine®. The other aims are to determine the factors which have an influence over the success or the failure of direct pulp capping.

Method : The patient's non-opposition is obtained after a loyal explanation of the study in order to collect clinical data, if a pulpal exposure (<2mm) happens on a vital tooth during decy excavation.

The operator registers the following data: age of the patient, type of the concerned tooth, volume of coronal pulp, surface of the pulp exposure, location, area and duration of pulp bleeding. An evaluation is realized 3 months later with the same clinical evaluation and a radiographic evaluation. If the pulp vitality is normal, the final coronal filling is then realized.

A statistical analysis will be performed to determine the success rate (binomial distribution with p=0.05). The predictive factors of success or failure will be analyzed with a logistic regression (with p=0.05).

ELIGIBILITY:
Inclusion Criteria:

* adult patients with a small pulp exposure (<2mm) created during decy removal on a vital tooth
* absence of spontaneous pain, of fistula, of swelling, of mobility, of periodontal enlargement, of resorption, of periapical pathosis, of furcation defect, on this tooth
* normal periodontal probing around this tooth
* cold vitality test : positive but non increased on this tooth

Exclusion Criteria:

* patient with at risk of endocarditis,
* patient with allergic reactions to a product used in the protocol,
* patient with a lack of oral hygiene,
* tooth with spontaneous pain, fistula, swelling, increased mobility, periodontal enlargement, resorption, periapical pathosis, furcation defect, pulpal necrosis, pulpal irreversible inflammation, excessive dental destruction, very abundant pulp bleeding, impossible set-up of the rubber dam
* tooth with a pulp exposure >2mm

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: adult patients with a small pulp exposure (<2mm) created during carie removal on a vital tooth
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-05-27 (Actual); Primary Completion 2016-12-02 (Actual); Study Completion 2016-12-02 (Actual)

PRIMARY OUTCOMES:
Treatment success | 3 months after the dental direct pulp capping
  Treatment success will be asses only if clinical AND radiographic examination are successful

CONTACTS AND LOCATIONS:
Locations (1):
- Chevalier, Brest, France